CLINICAL TRIAL: NCT01877772
Title: Trephination in Arthroscopic Cuff Repair: a Prospective Randomized Controlled
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Panam Clinic (Other); London Health Sciences Centre (Other); University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-0211
Record Dates: First submitted 2013-06-12; First posted 2013-06-14 (Estimated); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Rotator Cuff Tear
Keywords: cuff repair; arthroscopic; Trephination; Bone; cuff tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bone Trephination (Active Comparator): For the bone trephination, the wire will be advanced into the insertion site through the cortex and into the metaphyseal bone of proximal humerus.
  Interventions: Procedure: Bone Trephination; Procedure: Control
- Control (Active Comparator): The control group will undergo standard rotator cuff repair.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Bone Trephination — For the bone trephination, the wire will be advanced into the insertion site through the cortex and into the metaphyseal bone of proximal humerus.
  Arms: Bone Trephination
Procedure: Control — The control group will undergo standard rotator cuff repair.

SUMMARY:
This Clinical Trial is being conducted to study an adjunctive treatment for rotator cuff repair; bone trephination."Trephination" is a procedure that involves making small perforations in the bone that the tendon is repaired to.The rotator cuff is repaired by sewing the tendon down to the bone in the shoulder. Trephination is a new technique that is used in addition to the standard method of repairing the rotator cuff tendon. The control group will undergo the standard repair for rotator cuff tears.

It is the investigators' hypothesis that healing rates in patients who undergo bone trephination will be higher compared with surgery without trephination in arthroscopic rotator cuff repair at 24 months post-operatively.

DETAILED DESCRIPTION:
Rotator cuff repair carried out with current techniques has shown favourable results in terms of pain relief. However the re-tear rates remain high and are associated with significant morbidity in terms of functional outcome and shoulder strength. As rotator cuff disease becomes ever more prevalent with our aging population, it is imperative to determine if healing rates can be improved with autologous stem cell enhancement with pre-surgical preparation of the tendon insertion site through trephination. This trial is necessary both to provide optimal care of our patients, and to do so in a fiscally responsible fashion.

The primary outcome measure the re-tear rate as measured by ultrasound at 24 months post-operatively.

The secondary outcome measures are Western Ontario Rotator Cuff Index (WORC), Constant Score, and the American Shoulder and Elbow surgeons standardized assessment of shoulder function (ASES).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have failed standard non-surgical management of their rotator cuff tear, and who would benefit from a surgical repair of the cuff.

   Failed medical management will be defined as persistent pain and disability despite adequate standard non-operative management for 6 months. Medical management will be defined as:
   1. The use of drugs including analgesics and non-steroidal anti-inflammatory drugs
   2. Physiotherapy consisting of stretching, strengthening and local modalities (ultrasound, cryotherapy, etc)
   3. Activity modification
2. Imaging, and intra-operative findings confirming a full thickness tear of the rotator cuff.

Exclusion Criteria:

1. Characteristics of the cuff tear that render the cuff irrepairable:

   fatty infiltration in the muscles grade III (50%) or greater; superior subluxation of the humeral head; retraction of the cuff to the level of the glenoid rim.
2. Partial thickness cuff tears.
3. Significant shoulder comorbidities e.g. Bankart lesion, osteoarthritis
4. Previous surgery on affected shoulder e.g. Previous rotator cuff repair.
5. Isolated subscapularis tendon tears
6. Active joint or systemic infection
7. Significant muscle paralysis
8. Rotator cuff tear arthropathy
9. Charcot's arthropathy
10. Significant medical comorbidity that could alter the effectiveness of the surgical intervention (eg. Cervical radiculopathy, polymyalgia rheumatica)
11. Major medical illness (life expectancy less then 1 year or unacceptably high operative risk)
12. Unable to speak or read English/French
13. Psychiatric illness that precludes informed consent
14. Unwilling to be followed for 24 months
15. Advanced physiologic age

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
High-resolution ultrasound | 6 and 24 months post op
  High-resolution ultrasound will be used as the primary outcome measure to determine the re-tear rate at 6 and 24 months following repair. Ultrasound was chosen as it has been shown to have a high degree of accuracy for the diagnosis of rotator tears that is equivalent but less expensive than MRI.
  The interpretation of the high-resolution ultrasound is based on healing status and will be carried out by a trained MSK radiologist. Healing status will be documented at both 6 and 24 months as either completely healed, partially healed, or not healed. For tendons partially healed or not healed, the size of the defect will be compared with the size of the tear pre-operatively.

SECONDARY OUTCOMES:
Functional Outcome scores | baseline and 3, 6, 12, 18 and 24 months post op
  WORC, ASES and Constant

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lapner, MD, Principal Investigator — OHRI
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Zhao S, Liu G, Zhang D, Tang S. Intraoperative Channeling in Arthroscopic Rotator Cuff Repair: Letter to the Editor. Am J Sports Med. 2023 Jun;51(7):NP20. doi: 10.1177/03635465231169536. No abstract available. PMID 37259789
- [Derived] Lapner P, Bouliane M, Pollock JW, Coupal S, Sabri E, Hodgdon T, Old J, Mcilquham K, MacDonald P; CSES Investigators:; Stranges G, Berdusco R, Marsh J, Dubberley J, McRae S. Intraoperative Channeling in Arthroscopic Rotator Cuff Repair: A Multicenter Randomized Controlled Trial. Am J Sports Med. 2023 Feb;51(2):323-330. doi: 10.1177/03635465221138562. Epub 2022 Dec 1. PMID 36453726